CLINICAL TRIAL: NCT04246073
Title: Prospective Evaluation of Efficacy and Safety of Fondaparinux in Surgical Cancer Patients, Identification of the Most Relevant Risk Factors for Thromboembolism
Brief Title: Prospective Evaluation of Efficacy and Safety of Fondaparinux in Surgical Cancer Patients, Risk Factors for Thromboembolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Society of Surgical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 1787/11-2-2019
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-01

CONDITIONS: Cancer; Cancer Diagnosis; Thromboembolism
Keywords: Cancer; Cancer Diagnosis; Thromboembolism
MeSH Terms: conditions — Neoplasms; Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non interventional multi-centric study that will aim in evaluating the efficacy and safety of Fondaparinux in surgical cancer patients, identifying in parallel the most relevant and critical risk factors for Thromboembolism.

DETAILED DESCRIPTION:
Non interventional multi-centric study that will aim in evaluating the efficacy and safety of Fondaparinux in surgical cancer patients, identifying in parallel the most relevant and critical risk factors for Thromboembolism.

It is a cohort study, recruiting cancer patients over 18 years of age, who have been diagnosed with cancer for over a period of one year.

Exclusion criteria apply as well while all patients can withdraw their participation at any time point.

ELIGIBILITY:
Inclusion Criteria:

Upcoming surgery for newly diagnosed or potential cancer or relapse / metastasis of cancer that has been treated and diagnosed ≥ 1 year

Exclusion Criteria:

* Recent (<6 months) episode of venous thromboembolic disease (Deep vein thrombosis and / or pulmonary embolism and / or thrombosis in a rare location such as visceral or cerebral venous thrombosis)
* Pregnancy or pregnancy
* Patients on long-term anticoagulation for any reason (MKH, HMB or ABK, DOACs) at prophylactic or therapeutic dose, prior to enrollment in the study.
* Active haemorrhage, diagnosed hemorrhagic disorder, thrombocytopenia
* Ulcers or vasodilatations of the gastrointestinal tract
* Hemorrhagic stroke or surgery in the brain, spine or eye of the last trimester
* Bacterial endocarditis or other contraindication to the use of anticoagulant treatment
* Creatinine clearance <20mL / min
* Thrombolytic treatment or administration of dextran in the 2 days preceding administration of fondaparinux

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi centered, non interventional study with inclusion and exclusion criteria as described in the above section. Due to the fact that this is an observational study the results of all correlations will be carefully discussed and will used only for the evaluation of cases.Patients' participation in the study may be interrupted at any time.
  The reasons for the interruption could be as follows:
  1. Withdrawal of patient consent
  2. Incorrect enrollment in the study, ie the patient does not meet the inclusion / exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of incidents | One Year
  Observed number of incidents per cancer type
Number of bleeding episodes | One Year
  The incidence of bleeding episodes by type of cancer
Comparison of results/incidents among groups | One Year
  Results of treatment in subgroups of patients (for example patients with newly diagnosed cancer or potential cancer or relapse / metastasis of cancer that has been treated before and diagnosed ≥ 1 year)
Evaluation | One Year
  Evaluation of antithrombotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Karaitianos, Study Director — Hellenic Society of Surgical Oncology
Locations (1):
- Ioannis Karaitianos, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No